CLINICAL TRIAL: NCT03700073
Title: Correlation Between Physiological Cost Index and Health-related Quality of Life in Cerebral Palsy
Brief Title: Correlation Physiological Cost Index
Acronym: CPCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Eva Segura Ortí, Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-correlPCI
Record Dates: First submitted 2018-07-12; First posted 2018-10-09 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Cerebral Palsy
Keywords: physiological cost index; health-related quality of life; gait deviation index; gait analysis; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walk training plus virtual reality (Experimental): Experimental group (GTVR): The intervention consisted of treatment with the robotic CL1Walker gait training system in combination with virtual reality
  Interventions: Other: Experimental group (GTVR)
- Walk training (Active Comparator): Control group (GT): The intervention consisted of treatment with the robotic CL1Walker gait training system
  Interventions: Other: Control group (GT)

INTERVENTIONS:
Other: Experimental group (GTVR) — Gait training with a robotic system (CL1Walker) combined with immersion in a Virtual Reality program
  Arms: Walk training plus virtual reality
Other: Control group (GT) — Gait training with a robotic system (CL1Walker) alone.
  Arms: Walk training

SUMMARY:
Objective: To compare the efficacy of a gait training program using robotic assistance combined with virtual reality versus robotic assistance alone on energy expenditure in children with cerebral palsy.

Participants: Children with cerebral palsy levels II, III, IV, and V according to the Gross Motor Function Classification System (GMFCS), from different paediatric physiotherapy centres and schools in Valencia, Spain.

Intervention: Gait training using an inexpensive robotic gait training system (CL1Walker) and participation in a virtual reality game, Treasure Hunt (abbreviated here as ACT, from the Spanish A la Caza del Tesoro) in the experimental group (GTVR) and gait training using the same robotic gait training system without using virtual reality in the control group (GT).

Measurements: Assessment using the Physiological Cost Index (PCI) one week prior to and after the intervention. The intraclass correlation (ICC) replicability and the minimum detectable change (MDC) of the PCI.

DETAILED DESCRIPTION:
Design: Longitudinal, prospective, double blind study with two treatment groups and repeated measurements, controlled for the condition without virtual reality.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cerebral palsy
* Must be able to follow the instructions and participate in the game

Exclusion Criteria:

* Orthopaedic surgery in lower limb
* Botulinum toxin in lower limb

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Physiological cost index at 6 months | The test will be performed 6 month interval
  Index of gait efficiency trough Physiological Cost Index. It's a valuable indicator of gait efficiency in children with different Cerebral Palsy-related disability levels and it can predict their future level of societal activity and participation. To establish normal gait efficiency parameters, the Physiological Cost Index in children without disabilities is 0.4 with shoes and 0.38 barefoot .

CONTACTS AND LOCATIONS:
Overall Officials: Eva SEGURA-ORTÍ, PhD, Principal Investigator — Universidad CEU Cardenal Herrera, UCH CEU
Locations (1):
- Clínica de Fisioterapia Maite Montañana, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided